CLINICAL TRIAL: NCT04409795
Title: A Pilot Trial of Adding Oral Hypoglycemic Therapy to Insulin Treatment in Monogenic Variant Carriers of the Joslin 50-Year Medalist Study
Brief Title: Oral Hypoglycemic Therapy for Monogenic Variant Carriers of the Joslin Medalist Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-76
Record Dates: First submitted 2019-11-14; First posted 2020-06-01 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes; Monogenic Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HLA+ Group (Other): Participants who are high-risk HLA-DR3 and/or DR4 (+); monogenic variant (+) with rare exome variant ensemble learner (REVEL) score>0.75; and both glutamic acid decarboxylase (GAD65) and islet antigen (IA2) autoantibody (-)
  Interventions: Drug: Metformin Extended Release Oral Tablet; Drug: Sitagliptin
- HLA- Group (Other): Participants who are high-risk HLA-DR3 and DR4 (-); with known or yet unknown monogenic variants with REVEL score>0.75; and either GAD65 and IA2 autoantibody (-), or autoantibody (+) with titers close to the cutoff
  Interventions: Drug: Metformin Extended Release Oral Tablet; Drug: Sitagliptin

INTERVENTIONS:
Drug: Metformin Extended Release Oral Tablet — Initial oral hypoglycemic agent added to existing insulin treatment
Drug: Sitagliptin — Secondary oral hypoglycemic agent added to existing insulin treatment (for those who are intolerant to or unable to achieve glycemic targets with metformin)

SUMMARY:
The purpose of this study is to evaluate the efficacy of adding oral hypoglycemic agents (OHA) to existing insulin treatment in monogenic variant carriers of the Joslin 50-Year Medalist Study ("Medalists"), who are characterized by ≥50 years of insulin-dependent diabetes. Our primary objective is to evaluate whether the presence of human leukocyte antigen (HLA) high-risk alleles for diabetes (DR3 and/or DR4) can affect the effectiveness of OHA in these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Existing participants in the Joslin 50-Year Medalist Study
* Residing in the United States
* Capable of giving informed consent
* Known detectable C-peptide >0.05 ng/mL

Exclusion Criteria:

* Known diagnosis of cancer or active inflammatory disease such as rheumatoid arthritis, lupus, and inflammatory bowel disease
* Recent history of myocardial infarction, angioplasty, bypass surgery, heart failure, angina, stroke, or uncontrolled hypertension>160/100 during the past 3 months
* Known diagnosis of cognitive dysfunction, dementia or Alzheimer's disease
* Pre-existing liver disease or liver function tests (AST or ALT)>3x the upper limit of normal
* Pre-existing kidney disease (Chronic Kidney Disease Stage IV and below, or estimated glomerular filtration rate<45 mL/min/1.73 m2)
* Active use of immunosuppressants
* Recipients of prior islet cell or pancreas transplantation
* Inability to travel due to frailty or health reasons
* Donated blood within the previous two (2) months

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | 3 months and 6 months
  Change in HbA1c (%) between the two study groups

SECONDARY OUTCOMES:
Daily insulin dose | 3 months and 6 months
  Change in daily insulin dose (units/kg body weight) between the two study groups
Body mass index (BMI) | 3 months and 6 months
  Change in BMI between the two study groups. Weight and height will be combined to report BMI in kg/m^2.
C-peptide | 3 months and 6 months
  Change in C-peptide (ng/mL) between the two study groups
Total cholesterol | 3 months and 6 months
  Change in total cholesterol (mg/dL) between the two study groups
Low density lipoprotein (LDL)-cholesterol | 3 months and 6 months
  Change in LDL-cholesterol (mg/dL) between the two study groups
High density lipoprotein (HDL)-cholesterol | 3 months and 6 months
  Change in HDL-cholesterol (mg/dL) between the two study groups
Triglycerides | 3 months and 6 months
  Change in triglycerides (mg/dL) between the two study groups
Area under the plasma concentration versus time curve (AUC) of C-peptide | 6 months
  Change in AUC of C-peptide between the two study groups, as measured by the hyperglycemic/arginine clamp, at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: George L. King, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States